CLINICAL TRIAL: NCT06645431
Title: The Effect of Low Water Intake on Glucose Regulation Measured Using Continuous Glucose Monitoring in a Free-Living Environment
Brief Title: Effect of Low Water Intake on Glucose Regulation Measured Using Continuous Glucose Monitoring
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Responsible Party: Principal Investigator, Adam Seal, Principal Investigator, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 2023-230-CP
Record Dates: First submitted 2024-10-09; First posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Blood Glucose Concentration; Blood Glucose Self Monitoring
Keywords: Hydration; Blood Glucose; Water Intake; Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- High water intake (Experimental): For six days, participants will consume the NAM's recommended total water intake of 2.7 liters per day for women and 3.7 liters per day for men
  Interventions: Behavioral: Water Intake
- Low water intake (Active Comparator): For six days, participants will consume 0.7 liters per day for women and 1 liter per day for men.
  Interventions: Behavioral: Water Intake

INTERVENTIONS:
Behavioral: Water Intake — Previous studies have not observed blood glucose with adequate vs. low water intake in a free-living situation. The use of continuous glucose monitors allows this.

SUMMARY:
This clinical trial aims to learn if increasing water intake for five days can lower blood glucose in healthy, free-living individuals. The main question it aims to answer is whether increasing water intake will reduce daily blood glucose. Researchers will compare blood glucose when drinking adequate water to when the same individuals drink a low amount of water to see if blood glucose differs with water intake. Participants will be asked to drink a prescribed volume of water over two weeks while wearing a continuous glucose monitor and collecting two urine voids throughout each day.

DETAILED DESCRIPTION:
Twenty participants between 18 and 55 will be recruited from San Luis Obispo County using flyers, social media, local channels, and other online methods. Participants must be able to provide written and verbal consent to participate in the study. They must not currently be diagnosed with conditions, including, but not limited to, diabetes, pre-diabetes, pregnancy, and chronic illnesses. They must neither have received any surgery on their digestive tract nor be taking any oral contraceptives.

Surveys will be administered throughout the study consisting of validated surveys, which will be given out to participants via the encrypted data storage intermediary platform RedCap, which creates a unique identifier for each response to a survey and will be used to link responses across the study period for each participant. Participant's personal information will be password-protected and stored separately to be used for follow-up responses by Cal Poly investigators and research staff.

After participants complete the interest form and permit us to contact them, researchers will schedule the first visit to determine if participants are eligible, obtain consent for participation, and complete questionnaires assessing baseline physical activity, fluid intake, and diet. All participant visits will be scheduled through email or in person when the participant is on a prior visit to the laboratory. Any researcher contacting a participant for scheduling will use a Cal Poly email address and will only contact the participant's email provided in the interest form. Any scheduling email sent will follow the attached script. The second visit will occur in person and mark the start of the first six-day intervention. During this visit, researchers will place the continuous glucose monitor and Gene Active sensor and provide participants with resealable containers for urine collection and concealed bags to transport urine samples to the laboratory. Participants will be assigned to treatments in a counterbalanced fashion. For six days, participants will consume either the NAM's recommended total water intake of 2.7 liters per day for women and 3.7 liters per day for men (high water intake group, HWI) or 0.7 liters per day for women and 1 liter per day for men (low water intake group, LWI). Participants will be allowed to consume fluid ad libitum for four days. For the second six days, participants will consume either HWI or LWI, depending on the treatment completed in the first five days. Participants cannot drink fluids other than water and coffee/tea if requested. Water bottles will be provided with the prescribed amount of water for each day. Participants will collect two urine samples daily: a first-morning sample upon waking and an afternoon sample (2:00 PM-5:00 PM). Participants will deliver their urine containers to the laboratory every other day. Urine samples will be analyzed for specific gravity and volume.

In Redcap, participants will complete a daily mood disturbance questionnaire and a weekly solid food-to-water questionnaire. They will also complete daily food fluid intake questionnaires. This will include a urine void survey, where participants will track the number of times they urinated each day. Participants will be asked to align their food intake during the second five-day intervention with the same foods and amounts consumed during the first five-day intervention. During the four-day washout period, participants can eat however they want.

ELIGIBILITY:
Inclusion Criteria

* 18-55 years
* able to provide written and verbal consent

Exclusion Criteria:

* diabetes
* pre-diabetes
* pregnancy
* chronic illness
* No past surgery on the digestive tract
* taking any oral contraceptives

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-07-31 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Daily blood glucose | 14 days
  Area under the curve of daily blood glucose

SECONDARY OUTCOMES:
Urine specific gravity | 14 days
  Urine concentration

CONTACTS AND LOCATIONS:
Overall Officials: Adam D Seal, Ph.D., Principal Investigator — California Polytechnic State University-San Luis Obispo
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: No